CLINICAL TRIAL: NCT05234255
Title: Prospective Reliability and Validity Study of Urdu Version of Core Outcome Measure Index- Neck Scale
Brief Title: Urdu Version of Core Outcome Measure Index - Neck Scale: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00247
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Chronic Neck Pain
Keywords: Core Outcome Measure Index-NECK SCALE; Chronic Neck Pain; reliability; Validity; Urdu Version

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Purpose of this study is to culturally adapt and translate Core outcome measure index-Neck Scale into Urdu language as well as to investigate the reliability and validity in Pakistani population. Also check its correlation with Neck Disability-Index, Neck-pain and the disability-scale and Functional-Rating-Index.

DETAILED DESCRIPTION:
The English version of the Core outcome measure index-Neck Scale will be translated and culturally adapted Urdu Language. In Patients who suffer from Chronic-Neck Pain, Core outcome measure index-Neck Scale will be distributed among one hundred and twenty participants choose a convenience sampling technique based on pre-defined inclusion and exclusion criteria. To test intra and inter observation reliabilities for the final Core outcome measure index-Neck Scale, Neck-pain and the Disability Scale, Functional-Rating-Index and Neck-Disability-Index questionnaire will be filled on the same day, by two observers, and for the inter-observer's assessment, with an interval of 30 minute between the first and the second application. Third assessment will be carried out after 7 days by for intra-observer assessment. Data will be entered and analyzed using Statistical Package of Social Sciences Software Version 24. Internal consistency will be analyzed by using Cronbach-alpha-value. Test-retesting reliabilities will assesses using the intraclass correlation coefficient. Core outcome measure index-Neck Scale will be evaluated for content validities, construct validities, and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, including both Male and females (age ≥18).
* Participants with Chronic-Neck Pains lasting more than Three months Duration.
* Participants with sufficient Knowledge and understanding Urdu Language.

Exclusion Criteria:

* Participants with the history of Neck-pains due to deformity, existing central or peripheral nervous disorders and cervical spinal cord fracture were excluded.
* Participants having systematic diseases (tumor or articular Diseases).
* Participants with any Pertinent comorbidities, including heart attack, Cancer, cognitive Impairment's and mental disorders were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The people included in this study were chronic neck pain Individuals (Both Genders) Among Urdu speaking Pakistani population.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Core Outcome Measure Index-Neck | 1st day
  There are five domains in Core Outcome Measure Index - Neck Scale that describe pain, function, symptom specific well-being, quality of life and disability of the patient. In the summary of core outcome measure index-neck each domain score transformed to a 0-10 scale and these are then averaged to give a score of 0 to 10, higher score indicate the severity
Neck-Disability-Index | 1st day
  This questionnaire is used to assess the quality and functional activities of daily life. This assessment tool consists of 10 sub-items that includes pain, lifting activities, personally caring, working, headaches, sleep, drive and recreations. This questionnaire is intended to provide us with information on how your neck discomfort has impacted your capacity to function in daily life. The Neck-Disability-Index has enough support and applicability to maintain its position mostly used self-reporting measures for neck discomforts. The Neck-Disability-Index can be administered to assess a patient's current state as well as their progress during treatment.
Neck-pain Scale and the Disability Scale | 1st day
  The Neck-pain Scale and the Disabilities Scale is a composition index including about twenty items which measure the intensities of the Neck-pains and related disabilities. The 20-item checklist assesses neck mobility issues, the severity of neck discomforts the impact of neck traumas on the amount of hindrance everyday activity. The Neck-pain and Disability scale is an established tool for assessing results in individuals with neck discomfort It's simple to fill out for the participants, and it's simple to evaluate for the assessors. Its impact on professional, cultural, interpersonal, and practical areas of life, as well as the existence and severity of emotional components connected with it
Functional Rating Scale | 1st day
  The Functional Rating Index is a self report questionnaire that describes pain in the neck or back region. There are 10-Items in Functional Rating Index that used to measure pain and functional level. The 5-point scale is used to check the response of the patient, 0 on this scale represents no pain or functional ability and 4 represents sever or worse pain. The Functional Rating Index scores range from 0% to 100%, in which there is no disability at 0% and severe disability on 100%

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No